CLINICAL TRIAL: NCT02484807
Title: Effect of Pharmacologic Interaction Between Endothelin-Receptor-Antagonists and Phosphodiesterase-5 Inhibitors on Medication Serum Levels and Clinical Disease Status in Patients Wih Pulmonary Arterial Hypertension
Brief Title: Effect of Pharmacologic Interaction Between ERAs and PDE-5 Inhibitors on Medication Serum Levels and Clinical Disease Status in Patients With PAH
Acronym: EPIC
Status: Completed | Type: Observational
Sponsor: Heidelberg University (Other)
Responsible Party: Principal Investigator, Prof. Dr. med. Ekkehard Gruenig, Prof. Dr. med., Heidelberg University
Other Study IDs: EPIC-01
Record Dates: First submitted 2015-06-24; First posted 2015-06-30 (Estimated); Results first posted 2020-02-05 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (6):
- Bosentan + Sildenafil: Combination treatment with Bosentan + Sildenafil at baseline
  Interventions: Other: no intervention, only observation of different groups
- Bosentan + Tadalafil: Combination treatment with Bosentan + Tadalafil at baseline
  Interventions: Other: no intervention, only observation of different groups
- Ambrisentan + Sildenafil: Combination treatment with Ambrisentan + Sildenafil at baseline
  Interventions: Other: no intervention, only observation of different groups
- Ambrisentan + Tadalafil: Combination treatment with Ambrisentan + Tadalafil at baseline
  Interventions: Other: no intervention, only observation of different groups
- Macitentan + Sildenafil: Combination treatment with Macitentan + Sildenafil at baseline
  Interventions: Other: no intervention, only observation of different groups
- Macitentan + Tadalafil: Combination treatment with Macitentan + Tadalafil at baseline
  Interventions: Other: no intervention, only observation of different groups

INTERVENTIONS:
Other: no intervention, only observation of different groups

SUMMARY:
The development of disease-targeted medication for the treatment of pulmonary arterial hypertension (PAH) has significantly improved within the last years, leading to the development of 10 approved agents. Combination treatment with Endothelin-Receptor-Antagonists (ERA) and Phosphodiesterase-Type-5-Inibitors (PDE-5-Inhibitor) has become increasingly important for the treatment of PAH. In a recent press release, the results of the AMBITION study reported that an upfront combination treatment immediately after diagnosis leads to a delayed disease progression [4]. Thus, the question if there is a clinically relevant pharmaco-dynamic drug-drug interaction is of rising interest.

DETAILED DESCRIPTION:
Mechanisms of action Three ERAs have been approved for the treatment of PAH including the dual inhibitors Bosentan and Macitentan and the selective Endothelin Receptor type A inhibitor (ETA-Inhibitor) Ambrisentan. The dual antagonists inhibit both ETA- and the type B (ETB)-receptor, while the selective antagonist only affects the ETA-receptor [2]. The physiologic ligand of the receptors is Endothelin-1, which binds to the ETA-receptor and causes vasoconstriction and proliferation of the vascular smooth muscle cells. The binding to the ETB-receptor leads to an endogenous production of NO and prostacyclin in the endothelial cells.

PDE-5-Inhibitors include the two substances Sildenafil and Tadalafil. They inhibit the degradation of cyclic guanosine monophosphate (cGMPs), which triggers the vasodilative effect of endothelial NO.

Interaction There is evidence for the pharmacokinetic interaction (inhibition / induction of critical targets of drug metabolism and drug distribution) of both substance classes: the PDE-5-Inhibitors Sildenafil and Tadalafil are mainly eliminated in the liver by the hepatic enzyme Cytochrom-P450-Oxygenase type 3A4 (CYP3A4). The dual inhibitor Bosentan is both a substrate and an inductor of the Cytochrom-P450-Oxydase type 3A4 and type 2C9 [5,6].

It has already been shown in an in vivo-study, that simultaneous application of PDE-5-Inhibitors and Bosentan leads to a systemic reduction of the PDE-5-Inhibitor concentration of 40%, due to the CYP3A4-inducing effect of Bosentan [5]. Sildenafil, in contrast, leads to a decreased degradation of Bosentan in the liver with an approximately 50% increase in plasma leves. An anticipated result, especially when higher dosages of Sildenafil are applied, is the accumulation of Bosentan and reduction of Sildenafil levels.

A recent in vitro-study has shown that Tadalafil may also serve as CYP3A4-inductor, while this effect has not been detected for Sildenafil [7].

In contrast Macitentan which has been approved in 2013, has no clinically relevant CYP3A4-inducing effects. [8]. The in vitro-study has also detected a further interaction between ERAs and PDE-5-Inhibitors. Both PDE-5-Inhibitors Sildenafil and Tadalafil affect the transport molecules organic anion transporting polypeptides (OATPs), which are responsible for the hepatocellular intake of the dual ERA Bosentan. They also had a mild effect on the intake of Ambrisentan.

Sildenafil is a potent inhibitor of OATPs, whereas Tadalafil shows only minor inhibition of OATPs [7]. Both Sildenafil and Tadalafil significantly reduce the intracellular concentration of Bosentan in the liver, leading to a reduced degradation of Bosentan. For Ambrisentan this effect seemed to be less pronounced [7]. Consequently, this mechanisms of action lead to higher ERA-levels and to decreased PDE-5-Inhibitor plasma concentrations in patients receiving combination treatment. The most distinct interaction is expected for the combination of Sildenafil (PDE-5-Inhibitor) and Bosentan (ERA).

Up to now, the prevalence and role of this pharmacokinetic interaction for the clinical status and progression of the disease is not clear. Respective combination treatments have only been investigated in healthy male volunteers so far [5,9].

ELIGIBILITY:
Inclusion Criteria:

1. Men and women ≥ 18 years old
2. Diagnosis of PAH according to ESC/ERS-guidelines: patients with manifest pulmonary arterial hypertension, mean pulmonary arterial pressure ≥25mmHg, measured by right heart catheterization.
3. Combination treatment with ERA (Bosentan, Ambrisentan or Macitentan) and PDE-5-Inhibitor (Sildenafil or Tadalafil) for more than 3 months.

Exclusion Criteria:

1. Underage patients
2. Pregnancy or lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with pulmonary arterial hypertension receiving disease-targeted combination therapy
Sampling Method: Non-Probability Sample
Enrollment: 125 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ekkehard Grünig, MD, Principal Investigator — Thoraxclinic at the University Hospital Heidelberg
Locations (1):
- Centre for pulmonary hypertension, Thoraxclinic at the University Hospital Heidelberg, Heidelberg, Germany

REFERENCES:
- [Background] Galie N, Hoeper MM, Humbert M, Torbicki A, Vachiery JL, Barbera JA, Beghetti M, Corris P, Gaine S, Gibbs JS, Gomez-Sanchez MA, Jondeau G, Klepetko W, Opitz C, Peacock A, Rubin L, Zellweger M, Simonneau G; ESC Committee for Practice Guidelines (CPG). Guidelines for the diagnosis and treatment of pulmonary hypertension: the Task Force for the Diagnosis and Treatment of Pulmonary Hypertension of the European Society of Cardiology (ESC) and the European Respiratory Society (ERS), endorsed by the International Society of Heart and Lung Transplantation (ISHLT). Eur Heart J. 2009 Oct;30(20):2493-537. doi: 10.1093/eurheartj/ehp297. Epub 2009 Aug 27. No abstract available. PMID 19713419
- [Background] Humbert M, Sitbon O, Simonneau G. Treatment of pulmonary arterial hypertension. N Engl J Med. 2004 Sep 30;351(14):1425-36. doi: 10.1056/NEJMra040291. No abstract available. PMID 15459304
- [Background] Voelkel NF, Gomez-Arroyo J, Abbate A, Bogaard HJ, Nicolls MR. Pathobiology of pulmonary arterial hypertension and right ventricular failure. Eur Respir J. 2012 Dec;40(6):1555-65. doi: 10.1183/09031936.00046612. Epub 2012 Jun 27. PMID 22743666
- [Background] Wrishko RE, Dingemanse J, Yu A, Darstein C, Phillips DL, Mitchell MI. Pharmacokinetic interaction between tadalafil and bosentan in healthy male subjects. J Clin Pharmacol. 2008 May;48(5):610-8. doi: 10.1177/0091270008315315. Epub 2008 Feb 27. PMID 18305126
- [Background] Paul GA, Gibbs JS, Boobis AR, Abbas A, Wilkins MR. Bosentan decreases the plasma concentration of sildenafil when coprescribed in pulmonary hypertension. Br J Clin Pharmacol. 2005 Jul;60(1):107-12. doi: 10.1111/j.1365-2125.2005.02383.x. PMID 15963102
- [Background] Weiss J, Theile D, Spalwisz A, Burhenne J, Riedel KD, Haefeli WE. Influence of sildenafil and tadalafil on the enzyme- and transporter-inducing effects of bosentan and ambrisentan in LS180 cells. Biochem Pharmacol. 2013 Jan 15;85(2):265-73. doi: 10.1016/j.bcp.2012.11.020. Epub 2012 Dec 5. PMID 23219525
- [Background] Weiss J, Theile D, Ruppell MA, Speck T, Spalwisz A, Haefeli WE. Interaction profile of macitentan, a new non-selective endothelin-1 receptor antagonist, in vitro. Eur J Pharmacol. 2013 Feb 15;701(1-3):168-75. doi: 10.1016/j.ejphar.2013.01.010. Epub 2013 Jan 23. PMID 23353592
- [Background] Burgess G, Hoogkamer H, Collings L, Dingemanse J. Mutual pharmacokinetic interactions between steady-state bosentan and sildenafil. Eur J Clin Pharmacol. 2008 Jan;64(1):43-50. doi: 10.1007/s00228-007-0408-z. Epub 2007 Nov 27. PMID 18040672

RESULTS

PARTICIPANT FLOW:
Recruitment Details: March 2015 - September 2015
Groups:
- Bosentan + Sildenafil: Combination treatment with Bosentan + Sildenafil at baseline
  no intervention, only observation of different groups
- Bosentan + Tadalafil: Combination treatment with Bosentan + Tadalafil at baseline
  no intervention, only observation of different groups
- Ambrisentan + Sildenafil: Combination treatment with Ambrisentan + Sildenafil at baseline
  no intervention, only observation of different groups
- Ambrisentan + Tadalafil: Combination treatment with Ambrisentan + Tadalafil at baseline
  no intervention, only observation of different groups
- Macitentan + Sildenafil: Combination treatment with Macitentan + Sildenafil at baseline
  no intervention, only observation of different groups
- Macitentan + Tadalafil: Combination treatment with Macitentan + Tadalafil at baseline
  no intervention, only observation of different groups
Period: Overall Study
Arm/Group | Bosentan + Sildenafil | Bosentan + Tadalafil | Ambrisentan + Sildenafil | Ambrisentan + Tadalafil | Macitentan + Sildenafil | Macitentan + Tadalafil
Started | 39 | 7 | 19 | 21 | 33 | 6
Completed | 39 | 7 | 19 | 21 | 33 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bosentan + Sildenafil | Bosentan + Tadalafil | Ambrisentan + Sildenafil | Ambrisentan + Tadalafil | Macitentan + Sildenafil | Macitentan + Tadalafil | Total
Number analyzed (Participants) | 39 | 7 | 19 | 21 | 33 | 6 | 125
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 23 | 3 | 7 | 7 | 14 | 2 | 56
  >=65 years | 16 | 4 | 12 | 14 | 19 | 4 | 69
Age, Continuous [Mean (Standard Deviation); unit: years] | 56 (16) | 56 (18) | 61 (19) | 63 (13) | 65 (13) | 64 (21) | 61 (16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 5 | 15 | 12 | 19 | 4 | 84
  Male | 10 | 2 | 4 | 9 | 14 | 2 | 41
Region of Enrollment [Number; unit: participants]
  Germany | 39 | 7 | 19 | 21 | 33 | 6 | 125

OUTCOME MEASURES:

1. Primary Outcome: Characterisation of Medication Levels
Description: comparison of different combination treatment arms (mean ± standard deviation), measurement of endothelin receptor antagonist plasma concentrations and PDE-5I plasma concentrations, results given es multiple of the expected mean plasma concentration (MOM). Due to technical setup measurement of plasma concentrations of macitentan was not possible.
  The expected mean concentration ranges (MOM) refer to data extracted from published plasma concentration-time profiles measured during monotherapy with sildenafil, tadalafil, bosentan, and ambrisentan and served as comparative values. Each individually measured drug concentration was set in proportion to the expected mean concentration and expressed as a multiple of the expected mean (MoM), with values <1 denoting lower and values >1 higher values than the expected mean.
Time Frame: baseline vs. measurement after 3-6 months
Measure: Mean (Standard Deviation); unit: MOM
Arm/Group | Bosentan + Sildenafil | Bosentan + Tadalafil | Ambrisentan + Sildenafil | Ambrisentan + Tadalafil | Macitentan + Sildenafil | Macitentan + Tadalafil
Number analyzed (Participants) | 39 | 7 | 19 | 21 | 33 | 6
MOM
  ERA concentrations | 5.54 (3.24) | 2.18 (1.23) | 1.81 (0.82) | 1.53 (0.84) | NA (NA) — measurement of Macitentan Plasma concentrations not possible due to technical limitations | NA (NA) — measurement of Macitentan Plasma concentrations not possible due to technical limitations
  PDE-5I concentrations | 0.44 (0.42) | 0.89 (0.53) | 1.30 (0.97) | 1.67 (0.63) | 1.16 (0.87) | 1.59 (0.99)

2. Secondary Outcome: Impact of Medication Adjustment
Description: Change of medication serum levels after clinically indicated medication adaptation in patients who received Bosentan + Sildenafil in the beginning and changed the ERA to Macitentan
  1. change of mean levels ± standard deviation
  2. frequency of borderline medication serum levels or medication levels out of the therapeutic window The expected mean concentration ranges (MOM) refer to data extracted from published plasma concentration-time profiles measured during monotherapy with sildenafil, tadalafil, bosentan, and ambrisentan and served as comparative values. Each individually measured drug concentration was set in proportion to the expected mean concentration and expressed as a multiple of the expected mean (MoM), with values <1 denoting lower and values >1 higher values than the expected mean.
Time Frame: baseline vs. measurement 3-6 months after switch
Population: 20 of 39 patients receiving bosentan /sildenafil were switched to macitentan. sildenafil concentrations were compared before and after switch.
Measure: Mean (Standard Deviation); unit: MOM
Groups:
- Bosentan / Sildenafil Indicated for Therapy Switch: patients from bosentan/sildenafil group who showed unsatisfying clinical response to current therapy were switched from bosentan to macitentan. Plasma concentrations were controlled after change of ERA.
Arm/Group | Bosentan / Sildenafil Indicated for Therapy Switch
Number analyzed (Participants) | 20
MOM
  sildenafil concentrations before switch | 0.42 (0.32)
  sildenafil concentrations after switch | 1.59 (1.46)

3. Secondary Outcome: Clinical Relevance 6 Minute Walking Distance
Description: * Changes of medication levels after adjustment of combination therapy if clinically indicated
  * correlation with clinical routine parameters indicating clinical disease status
Time Frame: baseline vs. measurement 3-6 months after switch
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Bosentan / Sildenafil Indicated for Therapy Switch
Number analyzed (Participants) | 20
meters
  6 minute walking distance before switch | 396 (118)
  6 minute walking distance after switch | 436 (108)

4. Secondary Outcome: Clinical Relevance NTproBNP
Description: as for outcome 3
Time Frame: baseline vs. measurement after 3-6 months
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Bosentan / Sildenafil Indicated for Therapy Switch
Number analyzed (Participants) | 20
ng/ml
  NTproBNP before switch | 2204 (3823)
  NTproBNP after switch | 1181 (2899)

5. Secondary Outcome: Clinical Relevance Echocardiography Systolic Pulmonary Arterial Pressure (sPAP)
Description: as for outcome 3
Time Frame: baseline vs. measurement after 3-6 months
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Bosentan / Sildenafil Indicated for Therapy Switch
Number analyzed (Participants) | 20
mmHg
  sPAP before switch | 60.6 (21.4)
  sPAP after switch | 60.2 (20.0)

6. Secondary Outcome: Clinical Relevance Echocardiography Tricuspid Annular Plane Systolic Excursion (TAPSE)
Description: as for outcome 3
Time Frame: baseline vs. measurement after 3-6 months
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Bosentan / Sildenafil Indicated for Therapy Switch
Number analyzed (Participants) | 20
mm
  TAPSE before switch | 21.9 (5.4)
  TAPSE after switch | 21.5 (5.9)

7. Secondary Outcome: Clinical Relevance Blood Gas Analysis Oxygen Saturation
Description: as for outcome 3
Time Frame: baseline vs. measurement after 3-6 months
Measure: Mean (Standard Deviation); unit: % oxygen saturation
Arm/Group | Bosentan / Sildenafil Indicated for Therapy Switch
Number analyzed (Participants) | 20
% oxygen saturation
  oxygen saturation before switch | 92.2 (4)
  oxygen saturation after switch | 93.0 (4)

ADVERSE EVENTS:
Time Frame: 6 months
Description: this is a non-interventional, cross-sectional cohort study. All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed.
Arm/Group | Bosentan + Sildenafil | Bosentan + Tadalafil | Ambrisentan + Sildenafil | Ambrisentan + Tadalafil | Macitentan + Sildenafil | Macitentan + Tadalafil
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
small sample size. Due to the fact that currently no established therapeutic plasma concentration ranges exist, no conclusion can be drawn whether lower or higher concentrations lead to treatment failure or adverse events.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less